CLINICAL TRIAL: NCT03063242
Title: Sargramostim to Reverse Myeloid Dendritic Cell Deficiency
Brief Title: Sargramostim for Myeloid Dendritic Cell Deficiency
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient resources necessary for completion.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB201600815; OCR16461 (Other: University of Florida)
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Kidney Diseases; Kidney Transplant
Keywords: Sargramostim
MeSH Terms: conditions — Kidney Diseases | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Project I will be used to optimize the dosage and timing of sargramostim administration with regard to the primary and secondary outcomes. Thus, Project II and III treatment will only begin once all 5 Project I participants have completed treatment and the data have been analyzed to guide subsequent dosing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Project I: Healthy participants (Experimental): 5 healthy participants will be used to optimize the dosage and timing of sargramostim administration with regard to the primary and secondary outcomes. Blood samples will be drawn and analyzed for mDC levels.
  Interventions: Drug: Sargramostim; Biological: Blood samples
- Project II: Patients with CKD stage IV/V (Experimental): 5 Patients with CKD stage IV/V who are cytomegalovirus (CMV) seropositive with mean blood mDC levels <1.0x104/mL will receive sargramostim treatment once all 5 healthy participants have completed treatment and the data have been analyzed to guide subsequent dosing. Blood samples will be drawn and analyzed for mDC levels.
  Interventions: Drug: Sargramostim; Biological: Blood samples
- Project III: kidney transplant patients (Experimental): 5 Kidney transplant recipients who are CMV seropositive with neutropenia (defined as absolute neutrophil count <1.0 x103/mm3) and/or CMV viremia will receive sargramostim treatment once all 5 Project I participants have completed treatment and the data have been analyzed to guide subsequent dosing. Blood samples will be drawn and analyzed for mDC levels.
  Interventions: Drug: Sargramostim; Biological: Blood samples

INTERVENTIONS:
Drug: Sargramostim — Study participants (n=5 per project) will receive subcutaneous injection of sargramostim (6 ug/kg) daily until maximal mDC levels are achieved, as determined by a dose response curve.
  Other Names: Leukine®, GM-CSF
Biological: Blood samples — Blood samples will be drawn at baseline and during each subsequent visit

SUMMARY:
The study will determine whether administration of sargramostim will improve myeloid dendritic cell deficiency in various study groups, including healthy subjects and patients with chronic kidney disease, including those with kidney transplants.

DETAILED DESCRIPTION:
The overall objective of this project is to study the ability of sargramostim to enhance mDC level and function, including subsequent stimulation of T cell responses, in various human subjects with demonstrated myeloid dendritic cell (mDC) and T cell deficiency.

Single center nonrandomized trial with an interrupted time series design involving measures on blood samples from three separate populations before and after administration of sargramostim.

The objective is to determine the safety and dose response of sargramostim administration in healthy participants and in patients with chronic kidney disease (CKD) and kidney transplants.

Additionally to determine whether reversal of mDC/T cell deficiency by sargramostim results in augmented T cell responses in these three groups.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years < 80 years
* Absence of acute or chronic medical condition and taking no prescription medications (Project I)
* Stable native or transplant kidney function (Project II/III)

Exclusion Criteria:

* Age < 18 or > 80 years
* History of non-adherence to prescribed medications (Projects II and III)
* Active drug or heavy alcohol use (defined as > 4 drinks/day)
* Pregnancy or breast feeding
* Active infection (bacterial or viral) or clinically significant infections within the past three months (e.g. those requiring hospitalization, or as judged by the PI, except for CMV viremia in Project III)
* Active malignancy (with the exception of excised non-metastatic basal cell carcinoma or squamous cell carcinoma of the skin, or adequately treated pre-invasive cervical cancer in situ)
* Unstable cardiovascular status (angina, arrhythmias, congestive heart failure (CHF) etc…)
* History of liver disease (as defined by a diagnosis of uncompensated cirrhosis)
* History of lung disease (including moderate-severe Chronic Obstructive Pulmonary Disease (COPD), interstitial lung disease, or asthma)
* Known hypersensitivity to yeast-derived products
* Hemoglobin < 10 g/dL and hematocrit < 30%.
* Abnormal white blood cell count (WBC) count at baseline (< 3 or > 12 x 103 cells/mm3, except Project III)
* Treatment with WBC growth factors (G-CSF or GM-CSF) or immunosuppressive medications (tacrolimus, cyclosporine, mycophenolate, azathioprine, corticosteroids, chlorambucil, cyclophosphamide) within 4 weeks of study (erythropoiesis-stimulating agents will be allowed for Project II and immunosuppression for Project III)
* Treatment with lithium within 4 weeks of study
* History of arterial or venous thrombosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-17 (Actual)

PRIMARY OUTCOMES:
Change in peripheral blood mDC levels | Baseline to 2 weeks
  mDC levels to >2.0 x104 mDCs/mL, with the target level defined as levels at or above upper quartile values in healthy controls

SECONDARY OUTCOMES:
Proportion of patients with adverse events during the intervention. | Baseline to 2 weeks
Increase in T cell levels, mDC Interleukin (IL)-12 production, and interferon-gamma (IFN-y) production in QuantiFERON-CMV and QuantiFERON-Monitor assays after the intervention. | Baseline to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karl Womer, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No